CLINICAL TRIAL: NCT04673071
Title: Effectiveness and Safety of Thread Embedding Acupuncture for Drug Resistant Epilepsy: a Randomized Clinical Trial
Brief Title: Effectiveness and Safety of Thread Embedding Acupuncture for Drug Resistant Epilepsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Minh-An Thuy Le, Lecturer, Principle Investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 617/UMP-BOARD
Record Dates: First submitted 2020-12-07; First posted 2020-12-17 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Epilepsy, Drug Resistant; Acupuncture Therapy
Keywords: Drug resistant epilepsy; Thread embedding acupuncture
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Intervention Model Description: 2-arm parallel design, randomized, controlled, assessor-blinded, clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thread Embedding Acupuncture (TEA) (Active Comparator): TEA once a month for 4 months + AEDs
  Interventions: Other: Thread Embedding Acupuncture (TEA)
- Sham-TEA (STEA) (Sham Comparator): STEA once a month for 4 months + AEDs
  Interventions: Other: Sham-TEA (STEA)

INTERVENTIONS:
Other: Thread Embedding Acupuncture (TEA) — TEA in 1 month for 4 months The six TEA points used in this study are GV20, BL15, BL18, ST40, GV14 and GB34.
  Acupuncture point Procedure Baihui (GV20) oblique insertion toward nose, 3cm Both Xin Shu (BL15) perpendicular insertion, 3cm Both Gan Shu (BL18) perpendicular insertion, 3cm Both Fenglong (ST40) perpendicular insertion, 3cm Dazhui (GV14) perpendicular insertion, 3cm Both Yanglingquan (GB34) perpendicular insertion, 3cm
  Arms: Thread Embedding Acupuncture (TEA)
Other: Sham-TEA (STEA) — STEA in 1 month for 4 months All procedure of Sham-TEA group, including acupoints and size of TEA will be same as that of TEA group. However, thread-removed TEA will be used for STEA group instead of normal TEA, and removing procedure of thread will be performed aseptic and secretly for patient-blinding and prevention of infection.
  Arms: Sham-TEA (STEA)

SUMMARY:
Epilepsy is one of the most common neurological diseases all over the world. Currently, about 70 million people have epilepsy worldwide. In particular, more than 30% of epilepsy patients still have seizures even though they are treated with appropriate anti-epileptic drugs (AEDs). This number has remained unchanged even after more than 20 years with many new anti-epileptic drugs being introduced. According to International League Against Epilepsy (ILAE), drug-resistant epilepsy is defined when a patient does not achieve seizure-free the seizure with two optimal antiepileptic drugs. This clinical trial is designed to evaluate the effectiveness and safety of thread-embedding acupuncture (TEA) as palliative treatment of drug resistant epilepsy.

DETAILED DESCRIPTION:
The objectives of this clinical trial are twofold: the effectiveness of TEA is assessed by comparing the changes in the seizure control and quality of life at 5 months between 2 groups: the TEA + baseline AEDs group and the sham-TEA (STEA) + baseline AEDs group. Adverse events (AEs) that occur during the study will be investigated to evaluate the safety of TEA.

This study is investigated by the following hypotheses:

* TEA can increase the probability of becoming seizure free.
* TEA can reduce the frequency and duration of seizures.
* TEA can improve quality of life.
* TEA is associated with adverse effects.

This clinical trial will be performed as a 2-arm parallel design, randomized, controlled, assessor-blinded, clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* People with drug resistant epilepsy
* Volunteers who agree to participate and sign the Informed Consent Form, following a detailed explanation of clinical trials

Exclusion Criteria:

* Under epilepsy surgery
* Inappropriate condition for thread-embedding acupuncture due to skin disease (the skin of the acupuncture point is swollen, hot, and red) or hemostatic disorder (PT INR (international normalized ratio )> 2.0 or taking anticoagulant)
* Pregnant women or other inappropriate condition for thread-embedding acupuncture
* Other diseases that could affect or interfere with therapeutic outcomes, including body exhaustion, severe gastrointestinal disease, cardiovascular disease, hypertension, diabetes, renal disease, liver disease or thyroid disorder
* TEA within 6 months previous
* Psychiatric disorder currently undergoing treatment such as depression or schizophrenia
* Heavy drinking (more than 3 cups per day)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11-17 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Seizure freedom | 1 Month
  Percentage of seizure reduction in seizure frequency compared to baseline seizure frequency. Seizure frequency is recorded by the participants using seizure diary.
Quality of life (QOL) | 5 months
  Quality of life was recorded by QOLIE-31 (Quality of Life in Epilepsy) questionnaire The Quality of Life in Epilepsy Inventory (QOLIE-31) contains seven multi-item scales that tap the following health concepts: emotional well-being, social functioning, energy/fatigue, cognitive functioning, seizure worry, medication effects, and overall quality of life. The scoring procedure for the QOLIE-31 first converts the raw coded numeric values of items to 0-100 point scores, with higher converted scores always reflecting better quality of life.

SECONDARY OUTCOMES:
Seizure Severity | 3 months
  The National Hospital Seizure Severity Scale (NHS3) was recorded The scale is administered by a health professional during an interview with a patient and a witness to the seizures. It contains seven seizure-related factors and generates a score from 1 to 27. The higher score reflects the more severity of seizure.
Epileptiform discharges | 5 months
  Epileptiform discharges (ED) were recorded in Electroencephalograph (EEG). Epileptiform discharges are defined as generalized or focal polyspikes, polyspike-wave, spike-wave, sharp and sharp - wave occurring in the forms of a single discharge or a burst. The duration of discharges are from 20 - 200 milliseconds. The EDs are interpreted and numbers of ED are counted during a standard EEG by trained neurologists.

CONTACTS AND LOCATIONS:
Overall Officials: Dan V Nguyen, MD, Principal Investigator — University of Medicine and Pharmacy at HCMC
Locations (1):
- Nguyen Tri Phuong Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Demographic characteristic and outcome data will be shared
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 1 year after the trial finish and for 2 years

REFERENCES:
- [Background] Cheuk DK, Wong V. Acupuncture for epilepsy. Cochrane Database Syst Rev. 2014 May 7;2014(5):CD005062. doi: 10.1002/14651858.CD005062.pub4. PMID 24801225
- [Background] Chao D, Shen X, Xia Y. From Acupuncture to Interaction between delta-Opioid Receptors and Na (+) Channels: A Potential Pathway to Inhibit Epileptic Hyperexcitability. Evid Based Complement Alternat Med. 2013;2013:216016. doi: 10.1155/2013/216016. Epub 2013 Apr 3. PMID 23662118
- [Background] Kim E, Kim HS, Jung SY, Han CH, Kim YI. Efficacy and safety of polydioxanone thread embedded at specific acupoints for non-specific chronic neck pain: a study protocol for a randomized, subject-assessor-blinded, sham-controlled pilot trial. Trials. 2018 Dec 6;19(1):672. doi: 10.1186/s13063-018-3058-9. PMID 30522504
- [Result] J. Zhang, Y. Z. Li, and L. X. Zhuang (2006). Observation on therapeutic effect of 90 tonic-clonic epilepsy patients treated by catgut implantation therapy. Zhen Jiu Lin Chuang Za Zhi, vol. 22, no. 6, pp. 8-10, 2006
- [Result] Kloster R, Larsson PG, Lossius R, Nakken KO, Dahl R, Xiu-Ling X, Wen-Xin Z, Kinge E, Edna Rossberg. The effect of acupuncture in chronic intractable epilepsy. Seizure. 1999 May;8(3):170-4. doi: 10.1053/seiz.1999.0278. PMID 10356376
- [Result] Da-ke XUAN, Advances of the study on acupoint catgut-embedding for epilepsy in recent 10 years, World Journal of Acupuncture - Moxibustion, Volume 22, Issue 3, 2012, Pages 37-46, ISSN 1003-5257, https://doi.org/10.1016/S1003-5257(12)60039-7.